CLINICAL TRIAL: NCT05657314
Title: A Comparison of Two Pea Proteins on Amino Acid Absorption, GI Tolerance, Muscle Damage and Recovery
Brief Title: Effects of Pea Proteins on Muscle Damage and Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Center for Applied Health Sciences, LLC (Industry)
Collaborators: Biohm Health, LLC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: BIOHM-1221
Record Dates: First submitted 2022-12-10; First posted 2022-12-20 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Pea Proteins; Muscle Damage; Amino Acid Change

STUDY DESIGN:
Intervention Model Description: Subjects will take a daily protein supplement (e.g., 15 g of pea protein or 15 g of pea protein + probiotic blend) for 4 weeks, have a 1-week washout period (i.e. meaning they will not take either supplement), and then take the alternate protein supplement for an additional 4 weeks.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comparator (Active Comparator): 15 grams of pea protein dissolved in 12 ounces of water.
  Interventions: Dietary Supplement: Active Comparator
- Active (Experimental): 15 grams of pea protein + probiotic blend (1 billion CFU/capsule - blend of Lactobacillus rhamnosus, Lactobacillus acidophilus, Saccharomyces boulardii, and Bifidobacterium breve) dissolved in 12 ounces of water.
  Interventions: Dietary Supplement: Active Comparator

INTERVENTIONS:
Dietary Supplement: Active Comparator — Consists of 15 grams of pea protein

SUMMARY:
This study is a double-blind, randomized, placebo-controlled, crossover clinical trial of N=40 recreationally active men to be recruited a single investigational center in Ohio (i.e., The Center for Applied Health Sciences).

Subjects will take a daily protein supplement (e.g., 15 g of pea protein or 15 g of pea protein + probiotic blend) for 4 weeks, have a 1-week washout period (i.e. meaning they will not take either supplement), and then take the alternate protein supplement for an additional 4 weeks. Outcome variables include plasma amino acids, muscle damage, muscle recovery, and GI tolerance.

DETAILED DESCRIPTION:
This study is a double-blind, randomized, placebo-controlled, crossover clinical trial of N=40 recreationally active men to be recruited a single investigational center in Ohio (i.e., The Center for Applied Health Sciences).

Subjects will take a daily protein supplement (e.g., 15 g of pea protein or 15 g of pea protein + probiotic blend) for 4 weeks, have a 1-week washout period (i.e. meaning they will not take either supplement), and then take the alternate protein supplement for an additional 4 weeks.

Subjects will attend 6 study visits. During Visit 1, subjects will be screened for participation (i.e., medical history, physical exam, routine blood work, background baseline diet). During Visit 2, subjects will get their vitals measured and become randomized into a treatment group. During visits 3 and 5, subjects will get their blood drawn to measure plasma amino acid (AA) responses before and 30, 60, 90, 120, 180 min post-ingestion of their protein test beverage (i.e., pea protein vs. pea protein + probotic) followed by an exhaustive workout to induce single leg muscle damage. During visits 4 and 6, subjects will get their blood drawn to measure the extent of muscle damage and assess their recovery. Also, during visits 3-6 subjects will undergo subjective assessments [markers of recovery (Perceived Recovery Scale) and visual analog scales (VAS) to assess changes in perceived recovery, GI gas and bloating, fatigue, muscle soreness/tightness, mood, and energy] and lower body girth measurements.

Comprehensive side effect profile/ adverse event monitoring will take place throughout the study duration.

ELIGIBILITY:
Inclusion Criteria:

* Provide voluntary signed and dated informed consent.
* Be in good health as determined by medical history and routine blood chemistries.
* Age between the ages of 18 and 55 (inclusive).
* Body Mass Index of 18.5-29.9 (inclusive).
* Subject agrees to maintain existing dietary patterns throughout the study period apart from ingesting the provided treatment beverage.
* Subject is willing and able to comply with the study and supplement protocol.
* Subject agrees to abstain from alcohol, coffee, and caffeinated beverages 24 hours prior to testing on all study visits.
* Subject agrees to abstain from strenuous exercise 72 hours prior to testing on all study visits.
* Body weight of at least 120 pounds.
* Normotensive (seated, resting systolic blood pressure <140 mm Hg and diastolic blood pressure < 90 mm Hg. If the first measurement is slightly elevated above these limits, the subject will be given a brief (5 minute) rest period, and two more measurements will be taken. The average of all three measurements will be used to determine eligibility.
* Normal seated, resting heart rate (<90 per minute).
* Willing to duplicate their previous 24-hour and fast for 8 hours prior each study visit.

Exclusion Criteria:

* Individuals who have been diagnosed with liver, renal, cardiovascular, or other metabolic disease.
* Use of any dietary supplements which may confound the study or its endpoints, including creatine, BCAA, HMB, betaine, beta-alanine, etc.
* Use of any prescription medications (particularly antibiotics and/or anti-inflammatories), or probiotics within the past 2 months which may confound the study or its endpoints.
* Alcohol consumption (more than 2 standard alcoholic drinks per day or more than 10 drinks per week) or drug abuse or dependence.
* Smokers.
* Clinically significant abnormal laboratory results at screening.
* Known sensitivity to any ingredient in the test formulations as listed in the Nutrition Facts label.
* Individuals who are cognitively impaired and/or who are unable to give informed consent.
* Individuals with diabetes, asthma, chronic inflammatory conditions (e.g., rheumatoid arthritis, colitis, IBS/IBD, gout or fibromyalgia, Crohn's disease, ulcerative colitis, Lupus, HIV/AIDS, etc.).
* Other known gastrointestinal or metabolic diseases that might impact nutrient absorption or metabolism, e.g., short bowel syndrome, diarrheal illnesses, history of colon resection, gastro paresis, Inborn-Errors-of-Metabolism (such as PKU).
* Individuals with excessive caffeine intake (600mg/day).
* Subjects who take medication which may adversely affect the measured outcomes (i.e., testosterone or other anabolic steroids, corticosteroids or testosterone replacement therapy (ingestion, injection, or transdermal), diuretics, etc.)
* History of malignancy in the previous 5 years except for non-melanoma skin cancer (basal cell cancer or squamous cell cancer of the skin).
* Prior gastrointestinal bypass surgery (i.e., Lapband, etc.).
* Women
* Currently participating in another research study with an investigational product or have been in another research study in the past 30 days.
* Any other condition which in the Investigator's opinion may adversely affect the subject's ability to complete the study or its measures or which may pose significant risk to the subject.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-01-06 (Actual); Primary Completion 2022-10-06 (Actual); Study Completion 2022-10-06 (Actual)

PRIMARY OUTCOMES:
Plasma amino acids | Change from baseline to 4 weeks.
  Plasma amino acid responses before and 30, 60, 90, 120, 180 min post-ingestion of the test product.
Lactate dehydrogenase (LDH) | Change from baseline to 24 hours after acute exercise.
  Concentration of LDH in plasma.
Creatine kinase (CK) | Change from baseline to 24 hours after acute exercise.
  Concentration of CK in plasma.
Myoglobin | Change from baseline to 24 hours after acute exercise.
  Concentration of myoglobin in plasma.
Blood Urea Nitrogen (BUN) | Change from baseline to 24 hours after acute exercise.
  Concentration of BUN in plasma.
Mid thigh circumference | Change from baseline to 24 hours after acute exercise.
  Mid thigh circumference as measured using a tape measure.

SECONDARY OUTCOMES:
Gastro Intestinal Bloating | Change from baseline to 4 weeks.
  Gastro-intestinal bloating as measured by a 10 cm visual analogue scale, where higher values represent greater bloating.
Gastro Intestinal Flatulence | Change from baseline to 4 weeks.
  Gastro-intestinal flatulence (gas) as measured by a 10 cm visual analogue scale, where higher values represent greater gas.
Fatigue | Change from baseline to 4 weeks.
  Fatigue as measured by a 10 cm visual analogue scale, where higher values represent greater fatigue.
Muscle Soreness | Change from baseline to 24 hours after acute exercise.
  Fatigue as measured by a 10 cm visual analogue scale, where higher values represent greater fatigue.

CONTACTS AND LOCATIONS:
Locations (1):
- The Center for Applied Health Sciences, Canfield, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided